CLINICAL TRIAL: NCT03258840
Title: The Effect of EPA on the Serum Activities of Paraoxonase 1, Homocystein, Thiolactonase and Some Indicators of Vascular Inflammation and PON2 Gene Expression in PBMC Ofthe Patients With Type II Diabetes
Brief Title: EPA Supplementation on Vascular Inflammation, and Gene Expression of PON2 in Patients With Type II Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 15202
Record Dates: First submitted 2017-07-16; First posted 2017-08-23 (Actual); Last update posted 2017-08-23 (Actual); Status verified 2011-12

CONDITIONS: Diabetes Mellitus Type II
Keywords: EPA; Paraoxonase 1; Paraoxonase 2; Type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Eicosapentaenoic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPA placebo (Placebo Comparator): EPA- placebo softgel (Containing 2 g edible paraffin oil), 2 times/day, for 8 weeks
  Interventions: Dietary Supplement: EPA Placebo
- EPA supplement (Active Comparator): EPA supplement softgel (containing 2 g EPA per day), 2 times/day, for 8 weeks.
  Interventions: Dietary Supplement: EPA Supplement

INTERVENTIONS:
Dietary Supplement: EPA Supplement — EPA supplement, 4 × 500 mg softgel daily (2 g per day), 2 times a day, for 8 weeks.
  Other Names: Eicosapentaenoic acid
  Arms: EPA supplement
Dietary Supplement: EPA Placebo — EPA- placebo softgel (Containing 2 g edible paraffin oil), 4 × 500 mg softgel daily, 2 times a day, for 8 weeks.
  Arms: EPA placebo

SUMMARY:
The aim of this study is to determining of the effects of Eicosapentaenoic acid (EPA) supplementation on serum activities of Paraoxonase-1 and Homocystein thiolactonase, and serum levels of some indicators of vascular inflammation, and the gene expression of PON2 in the peripheral blood mononuclear cell (PBMC) in the patients with type II diabetes mellitus.

DETAILED DESCRIPTION:
The aim of this study is to determining of the effects of Eicosapentaenoic acid (EPA) supplementation on serum activities of Paraoxonase-1 and Homocystein thiolactonase and several indicators of vascular inflammation and the gene expression of PON2 in the peripheral blood mononuclear cell (PBMC) in the patients with type II diabetes mellitus. In this randomized, double-blind clinical trial, placebo-controlled, single-center, 36 men and women aged 35-50 years with type 2 diabetes are enrolled in the study from the Iranian Diabetes Association. After signing informed consent, all individuals complete a general information form. a 24-hour food recall for 3 days will be taken from the participants at the beginning and the end of the study,. Selected samples are randomly classified into 2 blocks of groups receiving supplement and placebo. Two groups will be classified (blocked) based on sex. The supplement group, will receive 2 g/day EPA for 8 weeks and the placebo group will also receive placebo (containing 2 g of edible paraffin) (similar in terms of color, shape and size). Patients are recommended to sustain their diets and medication dose (s) during the study and also advised to maintain a constant level of physical activity. Blood samples will be collected after 8-12 hours fasting and anthropocentric variables, biochemical parameters, target gene expression and physical activity before and after the trial will be measured.

ELIGIBILITY:
Inclusion criteria:

* Willingness to collaborate in the study
* aged 35-50 years
* having a history of at least 1 year of type 2 diabetes mellitus before the participation in the study based on FBS ≥126 mg/dl or 2hPG ≥200 mg/dl (2-hour plasma glucose),
* 25≤BMI<30 kg/m2

Exclusion criteria:

* pregnant and breastfeeding women
* using insulin, alcohol consumption, smoking and other drugs
* taking drugs (lipid-lowering, β-blockers, diuretics, estrogens, progesterones, vitamin supplements and ω-3 fatty acid supplements
* followers of the special diet
* history of diabetic retinopathy or diabetic nephropathy
* type 1 diabetes mellitus and other disorders
* any need to take insulin, change in the dose (s) and type of medication or physical activity

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | Change from Baseline at 8 weeks after the intervention
  Hemoglobin A1c (HbA1c) measurement by related kits according their protocols

SECONDARY OUTCOMES:
PON2 gene expression | Baseline, 8 weeks after the intervention
  measurement of paraoxonase-2(PON-2) gene expression using quantitative Real-time PCR
Systolic blood pressure | Change frome baseline at 8 weeks
  Systolic blood pressure changes measurement by manometer
Diastolic blood pressure | Change frome baseline at 8 weeks
  Diastolic blood pressure changes measurement by manometer
serum paraoxonase-1(PON-1) activity | Baseline, 8 weeks after the intervention
  serum paraoxonase-1(PON-1) activity by kit according related protocol
PON1/HDL-c Ratio | Baseline, 8 weeks after the intervention
  calculating the ratio after measurement of PON1 and HDL-c by related kits according their protocols
serum paraoxonase lactonase (PON-HCTLase) activity | Baseline, 8 weeks after the intervention
  measurement of paraoxonase lactonase (PON-HCTLase) activity by related kit according its protocol
HDL-c | Baseline, 8 weeks after the intervention
  high density lipoprotein- cholesterol (HDL-c) measurement by related kits according their protocols
FBS | Baseline, 8 weeks after the intervention
  Fasting blood sugar (FBS) measurement by related kits according their protocols
HDL2-c | Baseline, 8 weeks after the intervention
  high density lipoprotein 2- cholesterol (HDL2-c) measurement by related kits according their protocols
HDL3-c | Baseline, 8 weeks after the intervention
  high density lipoprotein 3- cholesterol (HDL3-c) measurement by related kits according their protocols
Serum apo B | Baseline, 8 weeks after the intervention
  Serum apo-protein B measurement by related kits according their protocols
Serum apo A-I | Baseline, 8 weeks after the intervention
  Serum apo-protein A-I measurement by related kits according their protocols
apo B/apo A-I Ratio | Baseline, 8 weeks after the intervention
  calculating the ratio after measurement of apo B and apo A-1 by related kits according their protocols
Serum methionine | Baseline, 8 weeks after the intervention
  measurement of serum levels of methionine by related kit according its protocol
Serum malondialdehyde (MDA) | Baseline, 8 weeks after the intervention
  measurement of serum levels of malondialdehyde (MDA)by related kit according its protocol
Serum homocysteine (Hcy) | Baseline, 8 weeks after the intervention
  measurement of serum levels of homocysteine (Hcy) by related kit according its protocol
Serum sE-Selectin | Baseline, 8 weeks after the intervention
  measurement of serum levels of soluble E-Selectin by related kit according its protocol
sVCAM-1 | Baseline, 8 weeks after the intervention
  measurement of serum levels of soluble Vascular cell adhesion molecule-1 (VCAM-1) by related kit according its protocol
Serum cysteine | Baseline, 8 weeks after the intervention
  measurement of serum levels of cysteine by related kit according its protocol
Serum Lpa | Baseline, 8 weeks after the intervention
  measurement of serum levels of lipoprotein-a (Lpa)by related kit according its protocol

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Hassan Golzari, Ph.D, Principal Investigator — Department of Nutrition & Biochemistry, School of Public Health, Tehran University of Medical Sciences (TUMS); Mahmoud Djallali, Ph.D, Study Chair — Department of Nutrition & Biochemistry, School of Public Health, Tehran University of Medical Sciences (TUMS); Saeed Hosseini, MD,Ph.D, Study Director — Department of Nutrition & Biochemistry, School of Public Health, Tehran University of Medical Sciences (TUMS)
Locations (1):
- Tehran University of Medical Sciences (TUMS), School of Nutritional Sciences and Dietetics, Department of Cellular and Molecular Nutrition, Tehran, Iran

REFERENCES:
- [Derived] Golzari MH, Javanbakht MH, Ghaedi E, Mohammadi H, Djalali M. Effect of Eicosapentaenoic Acid Supplementation on Paraoxonase 2 Gene Expression in Patients with Type 2 Diabetes Mellitus: a Randomized Double-blind Clinical Trial. Clin Nutr Res. 2019 Jan 28;8(1):17-27. doi: 10.7762/cnr.2019.8.1.17. eCollection 2019 Jan. PMID 30746344